CLINICAL TRIAL: NCT02212678
Title: Repeated-Dose Oral N-acetylcysteine for the Treatment of Parkinson's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: Parkinson's Disease Society of the United Kingdom (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1406M51207; 123269 (Other: FDA)
Record Dates: First submitted 2014-08-04; First posted 2014-08-08 (Estimated); Results first posted 2019-05-16 (Actual); Last update posted 2019-05-16 (Actual); Status verified 2019-04

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Acetylcysteine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- N-acetylcysteine (Experimental): Subjects will be provided 6000 mg/day of N-acetylcysteine (capsule) to be divided into 2 equal daily doses and taken orally for approximately 28 days
  Interventions: Drug: N-acetylcysteine capsule

INTERVENTIONS:
Drug: N-acetylcysteine capsule — N-acetylcysteine capsule
  Other Names: NAC

SUMMARY:
The investigators are interested in evaluating the use of oral N-acetylcysteine (NAC) as therapy for Parkinson's Disease (PD) and measuring changes in brain and blood chemistry.

DETAILED DESCRIPTION:
The investigators are interested in evaluating the use of oral N-acetylcysteine (NAC) as therapy for Parkinson's Disease (PD) and measuring changes in brain and blood chemistry. The investigators' hypothesis is that repeated oral dosing of NAC will result in increased brain and red blood cell GSH concentrations in individuals with Parkinson's disease (PD) and healthy controls. The specific aims are to 1.) measure plasma and blood (red blood cell) glutathione (GSH) and ratio of reduced GSH to oxidized glutathione (GSSG) in individuals with PD and healthy controls at baseline and after four weeks of repeated high doses of oral NAC (6000 mg/day) and 2) measure cortical GSH levels (as ascertained through MRS) in those with PD and healthy controls at baseline and four weeks during repeated high doses of oral NAC (6000 mg/day) simultaneously with Aim 1. This study will combine information from a medical history, a physical examination, and disease rating scales with results obtained using Magnetic Resonance Spectroscopy (MRS) brain scans and pharmacokinetic studies from blood samples. This research will require 2 visits, one at baseline and one after approximately 28 days of therapy. Participants will provide their medical history during the first visit, and undergo a physical examination and rating scale each visit (duration: 1 hour). The first visit including the brain scans and blood collection will require approximately 3 hours of time. The brain scan and pharmacokinetic studies for the second visit will require approximately 8 hours of time. In total the second visit will take roughly 9 hours.

ELIGIBILITY:
Inclusion Criteria:

1. All participants must be 18 years or older
2. All enrollees must understand and cooperate with requirements of the study in the opinion of the investigators and must be able to provide written informed consent
3. Individuals with medically stable Parkinson's disease (in the opinion of the investigator)
4. All participants must not have taken antioxidants NAC, glutathione, coenzyme Q-10, vitamin C, or vitamin E for 3 weeks prior to the study
5. Absence of dementia in all subjects

Exclusion Criteria:

1. Inability to undergo MRI scanning without sedation and other MRI counterindications, such as metal in the body (see section 7.3)
2. Medically unstable conditions as determined by the investigators
3. Pregnant or lactating or those women of child-bearing age that are not using acceptable forms of contraception
4. Diagnosis of asthma that is presently being treated with any medication, or past history of asthma/bronchospasm resulting in an emergency room visit, hospitalization or treatment
5. Unable to adhere to study protocol for whatever reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2014-09; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Tuite, MD, Principal Investigator — University of Minnesota; Lisa Coles, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | N-acetylcysteine
Started | 8
Completed | 7
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | N-acetylcysteine
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 71 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Glutathione (GSH) Brain Levels
Description: GSH levels in brain of all subjects at baseline and post-NAC (n-acetylcysteine) dosing as measured by magnetic resonance spectroscopy (MRS)
Time Frame: pre-dose and after approximately 28 days of treatment
Measure: Mean (Standard Deviation); unit: mM
Arm/Group | N-acetylcysteine
Number analyzed (Participants) | 7
mM
  Baseline | 0.93 (0.33)
  Post-NAC | 0.99 (0.35)

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | N-acetylcysteine
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 4/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | N-acetylcysteine (N=8)
indigestion (Gastrointestinal disorders) | 4
increased tremor (Nervous system disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No